CLINICAL TRIAL: NCT02835612
Title: Early Intervention Program for Preterm Infants and Their Parents: Establishing the Impact at 18 Months Corrected Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Bill and Melinda Gates Foundation (Other); Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 150606; 150606 (Registry Identifier: Program for preterm infants)
Record Dates: First submitted 2016-07-11; First posted 2016-07-18 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Complication of Prematurity

STUDY DESIGN:
Intervention Model Description: we followed the SPIRIT 2013 statement. The research was approved by the hospital research committee.
  When infants reached 48 postnatal hours, they are sequentially randomized to the Enhanced Developmental Intervention (EDI) or Intervention Group or Usual Care or Conventional group (CG) using block randomization in a computer system (http://biostat.mc.vanderbilt.edu/wiki/Main/BlockRandomizationWithRandomBlockSizes). After the randomization, the intervention was initiated on the 7th postnatal day in the NICU (Neonatal Intensive Care Unit)
Who Masked: Investigator, Outcomes Assessor
Masking Description: IN THE NICU, intervention group received skin-to-skin care performed by the mother (kangaroo care) plus tactile-kinesthetic stimulation, also performed by the mothers, beginning at randomization, and continuing until hospital discharge. Infants in the Conventional Group (CG) received kangaroo care according to the routine of the NICU. After hospital discharge, we provided the cognitive-motor home-based intervention for infants in the IG and a home-based support protocol for all caregivers and parents. The principal investigators and the outcomes assessors didnt have known about the group that allocated patients and families (masked)
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early stimulation (Experimental): skin-to skin care by mother (kangaroo care) plus massage therapy by mothers.
  Interventions: Other: Early stimulation
- Conventional care (Active Comparator): skin-to skin care by mother (kangaroo care).
  Interventions: Other: Conventional care

INTERVENTIONS:
Other: Early stimulation — Intervention Group: skin-to skin care by mother ( kangaroo care ) plus massage therapy by mothers. They will receive the tactile-kinesthetic stimulation by mothers from randomization until hospital discharge. Intervention performed exclusively by the mothers was based on studies regarding the application of skin stimulations and passive exercises in preterm infants
  Arms: Early stimulation
Other: Conventional care — skin-to skin care by mother, kangaroo care. Standard care, according to the routine care of the NICU.
  Arms: Conventional care

SUMMARY:
There are several intervention programs involving multisensory and motor stimulations such as, gym, auditory, visual, vestibular and tactile stimulations. We propose to study a continuous program of early intervention involving very preterm infants' families in their first 12 months of life taking the chance of their neuronal plasticity during this period. Preterm infants born in our institution will be included when they complete 48 hours after birth (first intervention). All preterm infants and their mothers will be followed during neonatal period and pre hospital discharge they will have a second intervention ( to measure parental bond ). After discharge they will be conducted to follow up program and we will divided all very low birth weight infants included in the study in two groups according previous randomization:

1. Standard care with motor, and cognition evaluation and intervention according to their needs
2. Program of early intervention with parents' orientation independently of f the standard evaluation and care that will be performed.

All phases of neurodevelopment will be evaluated, and the parents will be oriented to stimulate motor, language and cognition iteratively and continuously at home; this is a innovative method to improve very preterm neurodevelopment outcome.

Randomization: in neonatal period, preterm infants will be sequentially randomized when they completed 48 hours after birth in:

Group 1- conventional group (CG): standard care, according to the routine care of the NICU (skin-to skin care by mother, kangaroo care ).

Group 2- intervention group (IG): skin-to skin care by mother ( kangaroo care ) plus massage therapy by mothers. They will receive the tactile-kinesthetic stimulation by mothers from randomization until hospital discharge. Intervention performed exclusively by the mothers was based on studies regarding the application of skin stimulations and passive exercises in preterm infants.

Both groups will receive skin-to skin care by mother (Kangaroo Care) according to the routine care of the neonatal intensive care unit (NICU).

DETAILED DESCRIPTION:
The main Goal is to develop a program of early intervention for very preterm infants that allows families to apply it continuously at home. An additional objective of this research is to quantify the results of early stimulation on improvement of cognition and motor skills.

Introduction- Born prematurely (soon to born) and its consequences cause major impact on society and health indicators of population. According to the 2012 ''Born Too Soon: The Global Action Report on Preterm Birth'' of the World Health Organization, Brazil is ranked 10th among the countries with the highest number of preterm live births and 16th in deaths due to complications of prematurity. The data from 2012 indicate that approximately 3 million babies are born in Brazil each year, 350 000 of whom are born with less than 37 weeks of gestation, and born prematurity index is higher in the last three years, including preterm very low birth weight infants gestational age (GA) less than 32 weeks and birth weight less than 1500 grams). More than half of the preterm infants with birth weight less than 1500 grams born in public university centers of Brazilian Neonatal network Research at a gestational age of 23-33 weeks died or were discharged with severe pulmonary, neurological or ophthalmological complication.

Early intervention for high risk preterm infant must focus in the parents-infant relationship, environment and behavioral attitudes. It is possible that a care process modified by households is beneficial for neurodevelopment premature, both in the cognitive aspect as motor.

Background Preterm infants are high risk for delayed neurodevelopment. Early intervention programs for preterm infants that focus on development while the babies are still in the hospital and post discharge from the hospital, and into the community setting may have a greater impact on long-term morbidity as they are able to focus more on family factors and the home environment. Interventions that are aimed at enhancing the parent-infant relationship focus on sensitizing the families to infants cues and teach appropriate and timely response to the preterm infant's needs, possibly that early high-quality parent-infant or mother-infant interactions positively influence cognitive and social development in children. Despite of those evidences, the role of the family applying those programs at home is not well studied especially in social deprived environments.

The groups and randomization according previous information in summary. In the NICU both groups will receive skin-to skin care by mother (Kangaroo Care) according to the routine care of the NICU, The mothers will be instructed to perform one stage at a time, and will be supposed to end the sequence within 15 min, four times per day with an interval of 6 hours.The tactile stimulation will be performed on the cutaneous surface and the muscular area corresponding to the temporal, frontal, periorbital, nasal and perilabial regions of the face; the external side of the upper and lower limbs; and the soft parts of two or three fingers grouped will be passed gently with moderate pressure, up to three times in one direction and three times in the opposite direction. The kinesthetic stimulation will consist of passive exercises (flexion and extension) of upper and lower limbs, one limb at a time and up to three times at each articulation (wrist, elbow, ankle and knee); one of the hands supporting the stimulated limb and the other hand performing the movements.

To ensure a safe application of the intervention, mothers of the IG will be instructed to observe the newborns' tolerance signs, avoid excessive stimulations, keep the babies lying on their back, with stretched limbs close to the body, and perform the kinesthetic stimulation to one limb at a time. Researchers of our team will have regular meetings with mothers included in IG every 48 hours to assure that they are doing the intervention as instructed and to check the parental bond PARENTAL BONDING INSTRUMENT (PBI) will be applied by a professional blind to the group to which the child belong.

Follow up appointments, home visits and intervention during follow up program The systematic orientation program for early intervention will be according to developmental milestones, anticipating in a month evolutionary step acquisition of motor and / or cognitive expected for corrected age. In the first half of corrected age, the mother, father and / or corresponding caregivers receive simple guidelines to encourage large motor skills, fine and cognition.

The time of these activities must not exceed 15 minutes and must seem game.Three times / week (alternating with gross and fine motor stimulation).

We will be perform two orientations every three months for cognitive stimulation, fine and gross motor , totaling the 10 home visits promoting guidance and supervision sessions. Systematic orientations will be delivered to parents in all medical appointments at follow up clinic.

There will be home visits in order to evaluate the comprehension of the orientation and to be sure that the intervention has been done by families.

There will be a multidisciplinary team involved in the whole study and we will have a critical view of the intervention impact (final evaluation) in both; conventional and intervention groups.

The infants will be evaluated in relation to their motor, and cognitive neurodevelopment using AIMS and Bayley III scales between 12 and 18 months corrected age.

AIMS (Alberta Motor Infant Scale): a blinded physiotherapist will evaluate the children of both groups between 12 and 18 months with Alberta Infant Motor (AIMS) scale in all eligible patients.

A global evaluation will be performed at one year chronological age with Bayley and AIMS scales.

The evaluation will be conducted in the presence of parents or caregivers in a safe surface with room for the child move around during the evaluation. The examiner will interact with the child to encourage response, but physical facilitation of movement should be avoided. During the evaluation, they are punctuated behaviors more or less mature within the motor repertoire of the child in each position (supine, prone, sitting and standing). This repertoire is called "motor" window. All items priced within the window motor and the window motor to the previous items are scored. The evaluation of the end, the child will receive a score based on the sum of the items scored on each posture, called raw score. This score will be observed in a standardized chart to find the baby development percentile according to the chronological age or corrected. Percentiles instrument standards are: 5%, 10%, 25%, 50%, 75%. According to this percentile baby's development can be classified into three categories: normal or typical (percentile> 25%), suspicious (BSDI-III: Bayley Scales of Infant and Toddler Development third edition: The Bayley Scales of Infant and Toddler Development, Third Edition, will be used for assessment of neurodevelopment at 12 and 18 months' corrected age. The scales will be administered at the hospital clinic, on the same day of each follow-up visit, by a psychologist who was blinded to group allocation. Cognitive, motor, and language development will be considered normal if higher than 89; below average if 80 to 89; borderline if 70 to 79; and extremely low if less or equal 69. Examine all the facets of a young child's development according manual.

AIMS and Bayley Scales are recommended to use together and a different ages because false positives are common and therefore it is beneficial to follow-up children at high risk of motor impairment at more than one time point, or to use a combination of assessment tools.

If this program shows a good result it can be expanded for the whole preterm population in order to improve their neurodevelopment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born in our institution will be included when they complete 48 hours after birth

Exclusion Criteria:

* Congenital malformations

Ages: 48 Hours to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Change in neurodevelopmental outcome | 4 months, 8 months 12 months and 18 months corrected age,
  Bayley scales III version

SECONDARY OUTCOMES:
Mortality | During NICU hospitalization and follow up program (up to 18 months CA)
  Measure by death during hospital stay and the follow at first two years of life
neuromotor outcome | one year corrected age
  AIMS instrument
home environment and maternal practices | one year corrected age
  Affordance in the Home Environment for Motor Development - Infant Scale - AHEMD-IS; Daily Activities of Infant Scale - DAIS ; the Knowledge of Infant Development Inventory - KIDI adapted for Brazilian children
Child/Mother interactions | 12 months corrected age
  Interaction Rating Scale - IRS, an observational tool, was used to measure the child's social skills, caregiver's parenting skills, and mother/child interactions. IRS includes 70 items about behaviors and yields ten subscales; five subscales (25 items) focus on children's social skills (i.e., autonomy, responsiveness, empathy, motor regulation, and emotional regulation) and the other five subscales (45 dichotomous items) on caregiver's parenting skills (i.e., respect for autonomy development, respect for responsiveness development, respect for empathy development, respect for cognitive development, and respect for social-emotional development); as well as an overall score of synchronous interactions between mother and the child

OTHER OUTCOMES:
Parent-Led Early Intervention in Very Preterm Infants: Effect on Executive Function at School Age | At school age.
  The long-term effects of enhanced early intervention on the executive functions of children born preterm. Executive function will be evaluated using NEPSY-II subtests measuring auditory attention, inhibition, design fluency, and motor persistence.

CONTACTS AND LOCATIONS:
Overall Officials: Rita C Silveira, MD PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guinsburg R, de Almeida MF, de Castro JS, Silveira RC, Caldas JP, Fiori HH, do Vale MS, Abdallah VO, Cardoso LE, Alves Filho N, Moreira ME, Acquesta AL, Ferrari LS, Bentlin MR, Venzon PS, Goncalves Ferri WA, Meneses Jdo A, Diniz EM, Zanardi DM, Dos Santos CN, Bandeira Duarte JL, Rego MA. Death or survival with major morbidity in VLBW infants born at Brazilian neonatal research network centers. J Matern Fetal Neonatal Med. 2016 Mar;29(6):1005-9. doi: 10.3109/14767058.2015.1031740. Epub 2015 Apr 2. PMID 25812674
- [Result] Silveira RC, Filipouski GR, Goldstein DJ, O'Shea TM, Procianoy RS. Agreement between Bayley Scales second and third edition assessments of very low-birth-weight infants. Arch Pediatr Adolesc Med. 2012 Nov;166(11):1075-6. doi: 10.1001/archpediatrics.2012.732. No abstract available. PMID 23007841
- [Result] Procianoy RS, Mendes EW, Silveira RC. Massage therapy improves neurodevelopment outcome at two years corrected age for very low birth weight infants. Early Hum Dev. 2010 Jan;86(1):7-11. doi: 10.1016/j.earlhumdev.2009.12.001. Epub 2009 Dec 22. PMID 20022717
- [Result] Silveira RC, Valentini NC, O'Shea TM, Mendes EW, Froes G, Cauduro L, Panceri C, Fuentefria RN, Procianoy RS. Parent-Guided Developmental Intervention for Infants With Very Low Birth Weight: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2421896. doi: 10.1001/jamanetworkopen.2024.21896. PMID 39018071
- [Result] Silveira RC, Mendes EW, Fuentefria RN, Valentini NC, Procianoy RS. Early intervention program for very low birth weight preterm infants and their parents: a study protocol. BMC Pediatr. 2018 Aug 9;18(1):268. doi: 10.1186/s12887-018-1240-6. PMID 30092772
- [Derived] Tarouco ML, Procianoy RS, O'Shea TM, Silveira RC. Parent-Led Early Intervention in Very Preterm Infants and Executive Function at School Age: Secondary Analysis of a Randomized Clinical Trial. JAMA Pediatr. 2026 Jan 20:e255866. doi: 10.1001/jamapediatrics.2025.5866. Online ahead of print. PMID 41557341